CLINICAL TRIAL: NCT04632121
Title: Early Administration of Oral Nicorandil in ST Elevation Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Intervention: A Randomized Controlled Trial
Brief Title: Oral Nicorandil in ST Elevation Myocardial Infarction Patients Undergoing Primary Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ahmed Abdel Nasser Abdel Rady (Other)
Responsible Party: Sponsor-Investigator, Ahmed Abdel Nasser Abdel Rady, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Nicorandil in STEMI Patients
Record Dates: First submitted 2020-10-31; First posted 2020-11-17 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Nicorandil
MeSH Terms: interventions — Nicorandil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: will receive standard treatment + 20 mg nicorandil prior to PPCI, and then maintained on 20 mg b.i.d for 3 months .
  Interventions: Drug: Nicorandil 20 MG
- Group B: will be given standard treatment, without nicorandil loading or maintainance.

INTERVENTIONS:
Drug: Nicorandil 20 MG — Nicorandil is a nicotinamide ester that dilates peripheral and coronary resistance vessels via action on ATP-sensitive potassium channels and possesses a nitrate moiety that promotes systemic venous and coronary vasodilation. As a result of these dual actions, nicorandil reduces preload and afterload and results in an increase in coronary blood flow. In addition to these effects, nicorandil may have cardioprotective actions mediated through the activation of potassium channel
  Other Names: PCI
  Groups: Group A

SUMMARY:
* To study the effects of early oral administration of nicorandil in the setting of PPCI among STEMI patients on early angiographic, electrocardiographic, echocardiographic and hard clinical outcomes.
* To assess the possible benefits of nicorandil on myocardial reperfusion through LGE- CMR substudy after 3 months.

DETAILED DESCRIPTION:
Nicorandil is a nicotinamide ester that dilates peripheral and coronary resistance vessels via action on ATP-sensitive potassium channels and possesses a nitrate moiety that promotes systemic venous and coronary vasodilation. As a result of these dual actions, nicorandil reduces preload and afterload and results in an increase in coronary blood flow. In addition to these effects, nicorandil may have cardioprotective actions mediated through the activation of potassium channel .

Previous study on the effect of nicorandil on patients with stable angina has shown significant improvement in outcome due to a reduction in major coronary events.

Acute occlusion of the coronary artery in the STEMI patient subjects the myocardium supplied by that vessel to acute myocardial ischemia, thereby demarcating the area at risk (AAR) of potential MI, should the acute coronary occlusion be sustained or permanent. If the period of acute myocardial ischemia is prolonged (more than 20 minutes) a "wave front" of cardiomyocyte death begins in the subendocardium and extends transmurally over time toward the epicardium.

The deprivation of oxygen and nutrient supply results in a series of abrupt biochemical and metabolic changes within the myocardium. The absence of oxygen halts oxidative phosphorylation, leading to mitochondrial membrane depolarization, ATP depletion, and inhibition of myocardial contractile function.

Ischemia-Reperfusion injury (IRI) is defined as the paradoxical exacerbation of cellular dysfunction and death, following restoration of blood flow to previously ischemic tissues. Reestablishment of blood flow is essential to salvage ischemic tissues. However reperfusion itself paradoxically causes further damage, threatening function and viability of the organ.

Early intra-coronary administration of nicorandil has been shown to reduce the damage in the myocardial microcirculation caused by PPCI and the myocardial infarct size in patients with AMI .

Nicorandil prior to reperfusion was suggested to improve coronary flow. Furthermore, suppression of ventricular arrhythmia, and improvement of left ventricular function were demonstrated in patients who suffered from AMI and underwent primary PCI. But the definite clinical benefits of nicorandil were not found, which may be due to the small sample size of the selected studies .

Compared with intracoronary use alone, the intracoronary and peripheral intravenous use of nicorandil can better improve myocardial microcirculation and short-term prognosis .

Nicorandil use prior and post PCI could decrease the occurrence rate of ventricular arrhythmia in STEMI patients undergoing emergent PCI, and this effect might be related with reduced QTd and QTcd post medication .

Whether oral nicorandil, which is more widely available and more affordable, would have clinical benefits in terms of measures of reperfusion, and LV recovery post-STEMI, when administered in the early phase of STEMI is still questionable, and warrants further research.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI eligible for PPCI.

Exclusion Criteria:

* Patients undergoing other reperfusion strategies, including fibrinolysis, rescue PCI or pharmacoinvasive PCI.
* Patients presenting with Cardiogenic shock or symptomatic hypotension (BP< 90/60 mmHg)
* Patients who have contraindications for nicorandil e.g. advanced hepatic disease.
* Patients not consenting to the study protocol.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All STEMI patients undergoing primary PCI in Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Angiographic evidence of epicardial successful reperfusion | 1 day around PCI
  Angiographic evidence of epicardil successful reperfusion including; TIMI flow grade, and TIMI frame count.
Angiographic evidence of tissue-level successful reperfusion | 1 day around PCI
  Angiographic evidence of tissue-level successful reperfusion (Myocardial blush grade).

SECONDARY OUTCOMES:
Electrocardiographic measures of repolarization dispersion | after 90 minutes of PPCI
  Electrocardiographic measures of repolarization dispersion including; QTc, QTD, T-peak to T-end interval (Tp-Te), and its dispersion, and Tp-Te/QT ratio, as well as ST segment resolution at 90 minutes from reperfusion.
Echocardiographic measures of LV recovery | before discharge and at 3 months after index event.
  Echocardiographic measures of LV recovery including; 2-D left ventricular ejection fraction, left ventricle volumes, Mitral regurge severity, and wall motion score index.
Speckle tracking for global longitudinal strain of left ventricle | before discharge and at 3 months after index event
  2D- Left ventricle Global longitudinal strain by speckle tracking echocardiography (only 50 patients in each group)

REFERENCES:
- [Background] Pi SF, Liu YW, Li T, Wang Y, Zhou Q, Liu BJ, Peng WJ, Li X, Wang YY, Huang L. Effect of sequential nicorandil on myocardial microcirculation and short-term prognosis in acute myocardial infarction patients undergoing coronary intervention. J Thorac Dis. 2019 Mar;11(3):744-752. doi: 10.21037/jtd.2019.02.23. PMID 31019762
- [Background] Feng C, Han B, Liu Y, Wang L, Niu D, Lou M, Lu C. Effect of nicorandil administration on myocardial microcirculation during primary percutaneous coronary intervention in patients with acute myocardial infarction. Postepy Kardiol Interwencyjnej. 2018;14(1):26-31. doi: 10.5114/aic.2018.74352. Epub 2018 Mar 22. PMID 29743901
- [Result] Xu L, Wang L, Li K, Zhang Z, Sun H, Yang X. Nicorandil prior to primary percutaneous coronary intervention improves clinical outcomes in patients with acute myocardial infarction: a meta-analysis of randomized controlled trials. Drug Des Devel Ther. 2019 Apr 29;13:1389-1400. doi: 10.2147/DDDT.S195918. eCollection 2019. PMID 31118574
- [Result] Wu M, Huang Z, Xie H, Zhou Z. Nicorandil in patients with acute myocardial infarction undergoing primary percutaneous coronary intervention: a systematic review and meta-analysis. PLoS One. 2013 Oct 22;8(10):e78231. doi: 10.1371/journal.pone.0078231. eCollection 2013. PMID 24167609
- [Result] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415
- [Result] Allen DG, Xiao XH. Activity of the Na+/H+ exchanger contributes to cardiac damage following ischaemia and reperfusion. Clin Exp Pharmacol Physiol. 2000 Sep;27(9):727-33. doi: 10.1046/j.1440-1681.2000.03329.x. PMID 10972541
- [Result] IONA Study Group. Effect of nicorandil on coronary events in patients with stable angina: the Impact Of Nicorandil in Angina (IONA) randomised trial. Lancet. 2002 Apr 13;359(9314):1269-75. doi: 10.1016/S0140-6736(02)08265-X. PMID 11965271
- [Result] P. Channel, A. Triphosphate, M. Infarction, A. T. Sensitive, and P. Channel, "Nicorandil Nicorandil," 2018.